CLINICAL TRIAL: NCT01111656
Title: SWiss Atorvastatin and Interferon-Beta 1b Trial In Multiple Sclerosis - Follow up Study ("SWABIMS Follow Up-study")
Brief Title: Efficacy, Safety and Tolerability of Atorvastatin 40 mg in Patients With Relapsing-remitting Multiple Sclerosis Treated With Interferon-beta-1b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Viollier AG, Basel, Switzerland (Unknown); PharmaPart (Industry)
Responsible Party: Prof. H. Mattle, Department of Neurology, Inselspital, Bern University Hospital, and University of Bern, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75/07
Record Dates: First submitted 2010-03-15; First posted 2010-04-27 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multi-center; randomized; prospective; parallel-group; rater-blinded; RR-MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Interferon beta-1b 250ug subcutaneously every other day
  Interventions: Drug: Interferon beta-1b group
- 2 (Experimental): Interferon beta-1b 250ug subcutaneously every other day AND atorvastatin 40mg every day (oral)
  Interventions: Drug: Interferon beta-1b/Atorvastatin group

INTERVENTIONS:
Drug: Interferon beta-1b group — Patients receive interferon beta-1b 250ug subcutaneously every other day
  Arms: 1
Drug: Interferon beta-1b/Atorvastatin group — Patients receive interferon beta-1b 250ug subcutaneously every other day AND atorvastatin 40mg every day (oral)
  Arms: 2

SUMMARY:
The "SWiss Atorvastatin and Interferon-Beta 1b Trial In Multiple Sclerosis - Follow up Study" is the follow up study of the "SWiss Atorvastatin and Interferon Beta-1b Trial In Multiple Sclerosis (SWABIMS)" (see http://www.clinicaltrials.gov. Identifier: NCT00942591) SWABIMS evaluated the efficacy, safety and tolerability of atorvastatin 40 mg in addition to interferon-beta 1b compared to interferon-beta 1b monotherapy in patients with relapsing-remitting multiple sclerosis for 15 month. The SWABIMS Follow up study observes patients that finish the SWABIMS study for another 12 month with ongoing unchanged medication.

DETAILED DESCRIPTION:
Background

Multiple sclerosis is a chronic inflammatory autoimmune disease of the central nervous system. Statins are lipid-lowering drugs which inhibit the 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA-) reductase, which is the main regulatory enzyme of cholesterol biosynthesis. In recent years many studies have demonstrated, that statins have anti-inflammatory and immunomodulatory properties in addition to their lipid-lowering effects. Therefore, statins may have therapeutic potential in immune-mediated disorders such as multiple sclerosis. Studies in experimental allergic encephalomyelitis (EAE), the animal model for the human demyelinating disease multiple sclerosis, as well as smaller studies in patients with relapsing-remitting multiple sclerosis showed beneficial effect on the course of the disease. But there are also reports of negative impact of statins on multiple sclerosis. Therefore, bigger studies are needed to investigate the therapeutical potential of statins in multiple sclerosis.

Objective

To assess the efficacy, safety and tolerability of the combination of atorvastatin 40mg p.o. daily and interferon-beta 1b sc e.o.d compared to monotherapy with interferon-beta-1b sc e.o.d in patients with relapsing-remitting multiple sclerosis for 12 month after completing the SWABIMS study.

Methods

Multi-center, rater-blinded, parallel-group, two arm, randomized study. Patients with relapsing-remitting forms of MS, respecting all inclusion/exclusion criteria, were randomized in the SWABIMS study in two equal-size parallel arms after three months of treatment with interferon-beta 1b, receiving atorvastatin 40mg/d or not in addition to interferon-beta 1b for 12 month.

After successful completion of the study, patients were asked to participate in the "SWABIMS Follow up study" for another 12 month with ongoing medication.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of the SWABIMS study
* Written informed consent

Exclusion Criteria

* Any disease other than multiple sclerosis that would better explain the patient's signs and symptoms
* Secondary progressive MS
* Uncontrolled severe medical disorder
* Participation in any other studies

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with new lesions on T2-weighted images after 12 months of treatment | Month 0
Proportion of patients with new lesions on T2-weighted images after 12 months of treatment | Month 12

SECONDARY OUTCOMES:
Gd-enhancing lesions on T1-weighted images after 12 months of treatment. | Month 0
Total T2-hyperintense lesion volume (burden of disease, BOD) after 12 months of treatment. | Month 0
Cortical atrophy (changes in brain volume, changes in grey matter and white matter) on magnetic resonance imaging (MRI) after 12 months of treatment | Month 0
Clinical disease progression (Expanded Disability Status Scale [EDSS], Multiple Sclerosis Functional Composite [MSFC] ) | Month 0
Functional systems scores (of Expanded Disability Status Scale [EDSS] and Multiple Sclerosis Functional Composite [MSFC] ) | Month 0
Number of relapse-free patients after 12 months of treatment | Month 0
Relapse rate after 12 months of treatment | Month 0
Time to first relapse | Month 0
Gd-enhancing lesions on T1-weighted images after 12 months of treatment. | Month 12
Total T2-hyperintense lesion volume (burden of disease, BOD) after 12 months of treatment. | Month 12
Cortical atrophy (changes in brain volume, changes in grey matter and white matter) on magnetic resonance imaging (MRI)after 12 months of treatment | Month 12
Clinical disease progression (Expanded Disability Status Scale [EDSS] , Multiple Sclerosis Functional Composite [MSFC] ) | Month 12
Functional systems scores (of Expanded Disability Status Scale [EDSS] and Multiple Sclerosis Functional Composite [MSFC] ) | Month 12
Number of relapse-free patients after 12 months of treatment | Month 12
Relapse rate after 12 months of treatment | Month 12
Time of first relapse | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Mattle, Prof., Principal Investigator — Dep. of Neurology, Bern University Hospital
Locations (1):
- Department of Neurology, Bern University Hospital, and University of Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Kamm CP, Mattle HP; SWABIMS Study Group. SWiss Atorvastatin and interferon Beta-1b trial In Multiple Sclerosis (SWABIMS)--rationale, design and methodology. Trials. 2009 Dec 14;10:115. doi: 10.1186/1745-6215-10-115. PMID 20003436
- [Background] Youssef S, Stuve O, Patarroyo JC, Ruiz PJ, Radosevich JL, Hur EM, Bravo M, Mitchell DJ, Sobel RA, Steinman L, Zamvil SS. The HMG-CoA reductase inhibitor, atorvastatin, promotes a Th2 bias and reverses paralysis in central nervous system autoimmune disease. Nature. 2002 Nov 7;420(6911):78-84. doi: 10.1038/nature01158. PMID 12422218
- [Background] Kwak B, Mulhaupt F, Myit S, Mach F. Statins as a newly recognized type of immunomodulator. Nat Med. 2000 Dec;6(12):1399-402. doi: 10.1038/82219. PMID 11100127
- [Derived] Kamm CP, El-Koussy M, Humpert S, Findling O, Burren Y, Schwegler G, Donati F, Muller M, Muller F, Slotboom J, Kappos L, Naegelin Y, Mattle HP; SWABIMS Study Group. Atorvastatin added to interferon beta for relapsing multiple sclerosis: 12-month treatment extension of the randomized multicenter SWABIMS trial. PLoS One. 2014 Jan 30;9(1):e86663. doi: 10.1371/journal.pone.0086663. eCollection 2014. PMID 24497963